CLINICAL TRIAL: NCT05601557
Title: Research on the Clinical Characteristics and Key Diagnosis and Treatment Technology of Genetic and Metabolic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sujun Zheng (Other)
Responsible Party: Sponsor-Investigator, Sujun Zheng, Ethics Committee Member, Beijing YouAn Hospital
Organization: Beijing YouAn Hospital (Other)
Other Study IDs: LL-2022-048-K
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Diagnosis ， Treatment， Genetic and Metabolic Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- hyperbilirubinemia: Gilbert syndrome Crigler-Najjar syndrome Dubin-Johnson syndrome Rotor syndrome PFIC BIRC
  Interventions: Other: There is no intervention
- Wilson disease: Leipzig score system was used for diagnosis, and the total score ≥4 points could be confirmed. The total score of 3 is suspected diagnosis, which requires further examination. A total score of 2 or less is not considered for diagnosis.
  Interventions: Other: There is no intervention
- Hemochromatosis: ① clinical manifestations of extensive skin pigmentation, bronzing; Decline to disappearance of sexual function; Mild hepatosplenomegaly, may appear jaundice; The heart is enlarged; Pain and swelling mainly in metacarpophalangeal joints; Decreased glucose tolerance and increased blood glucose; ② Serum iron was significantly increased, serum transferrin was normal or decreased, transferrin saturation was significantly increased, often more than 62%, serum ferritin was significantly increased, often more than 500ug/L; (3)/HJV/HAMP TFR2 / SLC40A1 HFE gene mutation.
  Interventions: Other: There is no intervention
- Glycogen accumulation disease: According to different types, there may be the following manifestations, which need specific analysis. ① Clinical manifestations of abdominal distension, fasting hypoglycemia and other symptoms; ② Laboratory examination showed metabolic acidosis, hyperlactic acidemia, hyperuricemia and hyperlipidemia; ③ Abdominal CT showed enlarged liver volume; ④ Serum glucosidase activity decreased; (5) the GAA/G6PC/SLC374A/AGL/PYG/PHK gene mutations.
  Interventions: Other: There is no intervention
- Other types of inherited metabolic liver disease
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — The genotype of the patients was analyzed.

SUMMARY:
1. Establish a follow-up cohort of genetic and metabolic liver disease in The Chinese population, and carry out research on disease spectrum, clinical characteristics and personalized diagnosis and treatment to improve the level of diagnosis and treatment.
2. Establish a multidisciplinary collaborative diagnosis and treatment model of genetic metabolic liver disease, develop and promote diagnosis and treatment paths, and improve the diagnosis and treatment ability of genetic metabolic liver disease in Beijing and even the whole country.
3. Establish a new CRISPR gene diagnosis technology to realize fast and low-cost genetic testing.
4. Elucidating the genetic mutation spectrum of common genetic and metabolic liver disease in China is helpful to accurate gene diagnosis and functional research.
5. Study the genotype-phenotype, mutation and clinical outcome relationship and influencing factors of the common genetic and metabolic liver disease population in China, to guide the early diagnosis, early treatment and improve the prognosis.

ELIGIBILITY:
Inclusion Criteria:

Meet the diagnostic criteria of each disease.

Exclusion Criteria:

1. Co-infected with hepatitis B virus, hepatitis C virus and HIV;
2. Patients with liver fibrosis and cirrhosis caused by other causes;
3. Patients with alcoholic liver disease and autoimmune liver disease;
4. Liver malignancy has been suggested or confirmed by evidence;
5. Combined with other serious systemic diseases.

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inherited metabolic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
death | 5 years
  Death during the study was the outcome event

IPD SHARING:
Plan to Share IPD: No